CLINICAL TRIAL: NCT02244021
Title: A Pilot Phase II Study With BRENTUXIMAB VEDOTIN as Pre-ASCT Induction Therapy in Relapsed/Refractory Hodgkin's Lymphoma Patients Non Responding to IGEV Salvage Treatment
Brief Title: BRENTUXIMAB VEDOTIN as Pre-ASCT Induction Therapy in R/R HL Patients Non Responding to IGEV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fondazione Italiana Linfomi - ETS (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FIL_BRidge
Record Dates: First submitted 2014-09-10; First posted 2014-09-18 (Estimated); Last update posted 2018-02-09 (Actual); Status verified 2018-02

CONDITIONS: Relapsed/Refractory Hodgkin's Lymphoma
Keywords: HD; Hodgkin's Lymphoma; RELAPSED-REFRACTORY
MeSH Terms: conditions — Hodgkin Disease | interventions — Brentuximab Vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BRENTUXIMAB VEDOTIN (Experimental): 1 arm for all patients
  Interventions: Drug: BRENTUXIMAB VEDOTIN

INTERVENTIONS:
Drug: BRENTUXIMAB VEDOTIN — Patients with FDG-PET positive after IGEV will be treated with brentuximab vedotin as followed: 1.8 mg/kg every 3 weeks as a 30-minute outpatient IV infusion for a total of 4 cycles of treatment
  Growth factors may be used at the discretion of investigators but are not routinely advised.
  Patients with FDG-PET negative after brentuximab vedotin treatment will be addressed to high dose chemotherapy followed by ASCT.
  Other Names: SGN-35

SUMMARY:
A pilot phase II study with brentuximab vedotin as pre-ASCT induction therapy in relapsed/refractory Hodgkin's lymphoma patients non-responding to IGEV salvage treatment.

DETAILED DESCRIPTION:
Brentuximab vedotin emerged as active single-agent in the treatment of relapsed or refractory HL.

Some patients don't reach a complete response after salvage treatment with IGEV (ifosfamide, gemcitabine, vinorelbine) and remain PET positive so the idea is to treat this subset of patients with brentuximab vedotin with the aim of achieving a complete remission before transplant.

ELIGIBILITY:
Inclusion Criteria:

1. Classical Hodgkin Lymphoma according to the WHO classification
2. Histologically confirmed CD30+ HL at diagnosis
3. Patients at the first line salvage therapy
4. FDG-PET positivity after two cycles of IGEV treatment
5. PBPCs should have been collected after the first or the second IGEV cycle
6. Age≥ 18 years
7. ECOG PS of 0-2
8. Life expectancy > 6 months.
9. Written informed consent
10. Patients available for periodic blood sampling, study-related assessments and management of toxicity
11. Females of childbearing potential must have a negative β-HCG pregnancy test result (pregnancy test should be performed at screening an on day 1 of cycle 1 prior to brentuximab vedotin treatment).
12. Female patient is either post-menopausal for at least 1 year before the screening visit or surgically sterile or if of childbearing potential, agree to practice 2 effective methods of contraception, at the same time, from the time of signing the informed consent through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
13. Male patients, even if surgically sterilized, (i.e., status post vasectomy) agree to practice effective barrier contraception during the entire study period and through 6 months after the last dose of study drug, or agrees to completely abstain from heterosexual intercourse.
14. Required baseline laboratory data: Absolute neutrophil count ≥ 1500/µl, Platelet count ≥ 75.000/ µl, Haemoglobin must be ≥ 8 g/dL, Serum bilirubin ≤ 1.5 times ULN, Serum creatinine < 2.0 mg/dL and/or creatinine clearance or calculated creatinine clearance > 40 mL/minute, Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 times ULN

Exclusion Criteria:

1. Peripheral neuropathy > Grade 1
2. Histologic diagnosis different from Hodgkin Lymphoma
3. First line treatment with BEACOPP
4. Compressive symptoms caused by the presence of Lymphoma
5. Patients treated previously with any anti-CD30 antibody.
6. Known hypersensitivity to any recombinant proteins, murine proteins, or excipients contained in the brentuximab vedotin formulation.
7. Known human immunodeficiency virus (HIV) positive
8. Known hepatitis B surface antigen-positive, or known or suspected active hepatitis C infection
9. Diagnosed or treated for another malignancy within 3 years before the first dose or previously diagnosed with another malignancy and have evidence of residual disease. Patients with nonmelanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection.
10. Patients with known history of any of the following cardiovascular conditions:Myocardial infarction within 2 years of randomization, New York Heart Association (NYHA) Class III or IV heart failure, Evidence of current uncontrolled cardiovascular conditions, including cardiac arrhythmias, congestive heart failure (CHF), angina, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities, Recent evidence (within 6 months before first dose of study drug) of a left-ventricular ejection fraction <50%
11. Patients with known active viral, bacterial, or fungal infection requiring treatment with antimicrobial therapy within 2 weeks prior to the first dose of brentuximab vedotin.
12. Patients with known active Grade 3 or higher viral, bacterial, or fungal infection within 2 weeks prior to the first dose of brentuximab vedotin.
13. Patients with known cerebral/meningeal disease (HL or any other etiology), including signs or symptoms of Progressive Multifocal Leukoencephalopathy
14. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to protocol.
15. Symptomatic neurologic disease compromising normal activities of daily living or requiring medications.
16. Patients who are pregnant, or lactating and breastfeeding.
17. Patients that have not completed any prior treatment chemotherapy and/or other investigational agents within at least 5 half-lives of last dose of that prior treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2014-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Complete response (CR rate) | 1 year and half from the beginning of the study
  Complete response will be defined according to recently updated international criteria (Cheson 2007), assuming that a negative PET is defined by DEAUVILLE scores 1 and 2.

SECONDARY OUTCOMES:
PFS | 2 years and half from the beginning of the study
  Additional study endpoint is final response to Brentuximab vedotin followed by autologous stem cell transplantation (ASCT), in terms of progression free survival (PFS).
Neurotoxicity rate | 1 year half from the beginning of the study
  Neurotoxicity of any grade defined as National Cancer Institute Common Terminology Criteria for Adverse Events , version 4.03 (NCI CTCEA, 2010)
Duration of remission (DR) | 2 years and half from the beginning of the study
  Additional study endpoint is final response to Brentuximab vedotin followed by autologous stem cell transplantation (ASCT), in terms of duration of remission (DR).

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Michele Carella, Prof., Principal Investigator — Hematology Division, IRCCS AOU San Martino, Genova, Italy
Locations (7):
- Italy (7):
  - Istituto di Ematologia "L. & A. Seragnoli" , Policlinico S. Orsola Malpighi, Bologna
  - Ematologia, IRCCS AOU San Martino-IST, Genova
  - Ematologia Ospedale Vito Fazzi, Lecce
  - Ematologia e Unità BMT IRCCS Istituto Nazionale dei Tumori, Milan
  - Università degli Studi di Modena e Reggio Emilia, D.A.I di Medicina diagnostica clinica e sanità pubblica, AOU Policlinico, Modena
  - Dipartimento di Oncologia Medica ed Ematologia, Istituto Humanitas, Rozzano
  - SC Ematologia - Azienda Ospedaliera AO Città della Salute e della Scienza, Torino